CLINICAL TRIAL: NCT02495597
Title: Lung Clearance Index (LCI) and Bronchial Inflammation in Patients With Bronchiolitis Obliterans (BO)
Brief Title: LCI and Bronchial Inflammation in Patients With BO
Acronym: FRABO-02
Status: Completed | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Dr. med. Martin Rosewich, Principal Investigator, Johann Wolfgang Goethe University Hospital
Other Study IDs: EC 124/13
Record Dates: First submitted 2015-07-06; First posted 2015-07-13 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Bronchiolitis Obliterans
Keywords: bronchial inflammation; Bronchiolitis obliterans; Sputum; Blood; Inflammation; adaptive immune system; innate immune system
MeSH Terms: conditions — Bronchiolitis Obliterans; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, sputum cells, sputum supernatans
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Subject-Group: Patients suffering from doctors diagnosed bronchiolitis obliterans
  Interventions: Other: no intervention - just observational
- Control Group: age- and sex matched to subject-group
  Interventions: Other: no intervention - just observational

INTERVENTIONS:
Other: no intervention - just observational

SUMMARY:
The investigators here compare lung function parameters (RV, RV/TLC and FEF75) with the results of the Lung Clearance index (LCI) . Further this study evaluates bronchial inflammatory markers in 20 patients with bronchiolitis obliterans at the age of 6 to 28 years compared with an age- and sex-matched control group. The investigators will perform a pulmonary function test (body plethysmography with DLCO) and compare the results with the LCI. Further we will measure the fraction of exhaled nitric oxide (FeNO) and draw a blood sample to determine the level of systemic inflammation. Finally induced sputum is collected and a cell count is performed, and cells and supernatants are analyzed for inflammatory markers. This study will set baseline markers for future interventional studies.

DETAILED DESCRIPTION:
The purpose of this study is to compare lung function values with the Lung clearance index of 20 Patients with Bronchiolitis obliterans aged between 6 up to 28 years. Further we aim to compare the bronchial Inflammation between the patients and a reference group with similar age conditions to determine possible outcome-parameters for following interventional studies.

The sputum samples will be processed and quantitatively analyzed to get a profile of the cytological composition.

(Sputum and serum samples are analyzed by quantitative real-time polymerase chain reaction (PCR) (qRT-PCR) and by cytometric bead assay (CBA).)

Methods and Work Programme:

* Measurement of nitric oxide in expired air (FeNO)
* Lung function testing with spirometry and body plethysmography
* Lung clearance index (LCI)
* Bronchodilation
* Blood test: blood count, CRP, RAST, serum inflammatory mediators, (genetic markers of the non-specific pulmonary defense system)
* Induced sputum for inflammatory mediators and microbiological investigations

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* between 6 and 28 years of age
* Known Bronchiolitis obliterans

  * no Bronchiolitis obliterans(depending on the study group)
* Ability to perform lung function tests and inhalation

Exclusion Criteria:

* Acute illness with systemic or bronchial inflammation
* every chronic condition or infection (eg HIV, tuberculosis, malignancy)
* pregnancy
* known alcohol and/ or drug abuse
* Inability to understand the extent and scope of the study
* Participation in another study

Ages: 6 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients suffering from Bronchiolitis obliterans and controls
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2013-04; Primary Completion 2013-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
LCI compared to RV/TLC%-pred. | during Visit 1 (single day, single observation)
  Correlation of these lung function Parameters in patients with BO compared to healthy controls

SECONDARY OUTCOMES:
change of sputum cell count over time (percentage of neutrophils) | during Visit 1 (single day, single observation)
  induced sputum will be analyzed for different cellular components such as alveolar macrophages, neutrophils, lymphocytes and others. Epithelial cells will be excluded
Comparison of low CrP | during Visit 1 (single day, single observation)
  serum parameter for systemic inflammation
FVC (%-pred.) | during Visit 1 (single day, single observation)
  To compare FVC (%-pred.)of patients suffering from BO with FVC (%-pred.)of a healthy control group
FEV1 (%-pred.) | during Visit 1 (single day, single observation)
  To compare FEV1 (%-pred.)of patients suffering from BO withFEV1 (%-pred.)of a healthy control group
Tiffeneau-Index | during Visit 1 (single day, single observation)
  To compare Tiffeneau-Index of patients suffering from BO with Tiffeneau-Index of a healthy control group
sRtot (%-pred.) | during Visit 1 (single day, single observation)
  To compare sRtot (%-pred.) of patients suffering from BO with sRtot (%-pred.) of a healthy control group
RV/TLC (%-pred.) | during Visit 1 (single day, single observation)
  To compare RV/TLC (%-pred.) of patients suffering from BO with RV/TLC (%-pred.) of a healthy control group
IL-6 (pg/ml) | during Visit 1 (single day, single observation)
  comparing IL-6 in Serum of patients with BO with healthy controls
IL-8 (pg/ml) | during Visit 1 (single day, single observation)1
  comparing IL-8 in Serum of patients with BO with healthy controls
IL-17 (pg/ml) | during Visit 1 (single day, single observation)
  comparing IL-17 in Serum of patients with BO with healthy controls
IL-6 (mRNA delta-delta-ct) | during Visit 1 (single day, single observation)
  compare IL-6 mRNA in Sputum cells of patients with BO with healthy controls
IL-8 (mRNA delta-delta-ct) | during Visit 1
  compare IL-8 mRNA in Sputum cells of patients with BO with healthy controls
IL-17 (mRNA delta-delta-ct) | during Visit 1 (single day, single observation)
  compare IL-17 mRNA in Sputum cells of patients with BO with healthy controls
Percentage of FOXP3 positive cells in Sputum | during Visit 1 (single day, single observation)
  compare percentage of FOXP3 positive cells in Sputum cells of patients with BO with healthy controls

CONTACTS AND LOCATIONS:
Overall Officials: Martin Rosewich, MD, Principal Investigator — Johann Wolfgang Goethe University Hospital
Locations (1):
- Children's Hospital, Goethe-University, Frankfurt am Main, Hesse, Germany

REFERENCES:
- See also: Kurland G, Michelson P. Bronchiolitis obliterans in children. Pediatr Pulmonol. 2005 Mar;39(3):193-208. Review — http://www.ncbi.nlm.nih.gov/pubmed/15635614
- See also: Smith KJ, Fan LL. Insights into post-infectious bronchiolitis obliterans in children. Thorax. 2006 Jun;61(6):462-3. — http://www.ncbi.nlm.nih.gov/pubmed/16738042
- See also: Pichler M, Herrmann G, Schmidt H, Ahrens P, Zielen S. Persistent adenoviral infection and chronic obstructive bronchitis in children: is there a link? Pediatr Pulmonol. 2001 Nov;32(5):367-71. — http://www.ncbi.nlm.nih.gov/pubmed/11596161
- See also: Pichler MN, Reichenbach J, Schmidt H, Herrmann G, Zielen S. Severe adenovirus bronchiolitis in children. Acta Paediatr. 2000 Nov;89(11):1387-9. — http://www.ncbi.nlm.nih.gov/pubmed/11106056